CLINICAL TRIAL: NCT03914131
Title: To Evaluate the Efficacy and Safety of Xinnaoning Capsule in Treating Chronic Stable Angina Pectoris (Qi Stagnation and Blood Stasis Syndrome) : a Randomized, Double-blind, Parallel Controlled, Multi-center Clinical Study
Brief Title: Clinical Trial Scheme of Xinnaoning Capsule
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Duheng for Drug Evaluation and Research Co., Ltd. (DDER) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DHZD-XNNJN-001
Record Dates: First submitted 2019-03-28; First posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Chronic Stable Angina Pectoris; Qi Stagnation and Blood Stasis Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): Introduction period: 2 weeks, time window (±2 days). Dosage regimen: Take Xinnaoning Capsule Simulator 3 tablets per time, 3 times per day, orally, after meals.
  The treatment period: 12 weeks, time window (±4 days). Dosage regimen:Take Xinnaoning Capsule 3 tablets per time, 3 times per day, orally, after meals.
  Dosage form:Capsule
  Interventions: Drug: Xinnaoning Capsule; Other: Xinnaoning Capsule Simulator
- control group (Placebo Comparator): Introduction period: 2 weeks, time window (±2 days). Dosage regimen: Take Xinnaoning Capsule Simulator 3 tablets per time, 3 times per day, orally, after meals.
  The treatment period: 12 weeks, time window (±4 days). Dosage regimen:Take Xinnaoning Capsule Simulator 3 tablets per time, 3 times per day, orally, after meals.
  Dosage form:Capsule
  Interventions: Other: Xinnaoning Capsule Simulator

INTERVENTIONS:
Drug: Xinnaoning Capsule — Xinnaoning Capsule used in study group(treatment period) is the true drug that the investigators are to evaluate.
  Other Names: Xinnaoning
  Arms: study group
Other: Xinnaoning Capsule Simulator — Xinnaoning Capsule Simulator used in control group and introduction period(both groups) is the placebo to reduce the risk of bias.
  Other Names: placebo

SUMMARY:
This study is a randomized, double-blind, parallel-controlled, multicenter clinical study to evaluate the efficacy and safety of Xinnaoning capsule in the treatment of chronic stable angina pectoris (Qi stagnation and blood stasis syndrome).

DETAILED DESCRIPTION:
Coronary heart disease angina pectoris is a kind of heart disease caused by myocardial ischemia and anoxia caused by coronary atherosclerosis. It belongs to the category of "chest obstruction" and "heartache" in traditional Chinese medicine. One of its common pathogenesis is stagnation of Qi and blood stasis, blockage of blood vessels, so it should be treated by activating blood circulation and removing blood stasis, dredging channels and collaterals, as well as tranquilizing Qi and tranquilizing spirit, in order to achieve the goal of blood stasis to remove new life and nourish the blood vessels of viscera and viscera. Xinnaoning Capsule (Chinese medicine approved character: Z20025697) is produced by Guizhou Jingcheng Pharmaceutical Co., Ltd. It has the functions of activating blood circulation, promoting Qi circulation, dredging collaterals and relieving pain.Xinnaoning Capsule has not had any adverse reactions for many years after it was put on the market. In this study, a randomized, double-blind, placebo-controlled, multi-center, efficacy test design was used to evaluate the efficacy and safety of Xinnaoning Capsule in the treatment of chronic stable angina pectoris (Qi stagnation and blood stasis syndrome) .

ELIGIBILITY:
Inclusion Criteria:

* Refer to the Guidelines for Diagnosis and Treatment of Chronic Stable Angina issued by the Chinese Medical Association in 2007, 2012ACP/ACCF/AHA/AATS/PCNA/STS (Guidelines for Diagnosis and Management of Stable Ischemic Heart Disease: American Heart Foundation/American Heart Association/American Medical Association/American Thoracic Surgery Association/American Association for Cardiovascular Preventive Nursing/American Association for Cardiovascular Angiography and Intervention/American Thoracic Association The Diagnosis of Stable Ischemic Heart Disease: Guidelines for Clinical Practice, Guidelines for the Management of Stable Coronary Artery Diseases in 2013 ESC, which can diagnose coronary heart disease in accordance with any of the following:

  1. Has a clear history of old myocardial infarction, or PCI history, or bypass history
  2. Coronary angiography (results indicate at least one coronary artery stenosis with stenosis (>50%) or coronary CTA suggests stenosis with stenosis (>50%)
* Those who met the diagnostic criteria of chronic stable angina pectoris: those who had a history of angina pectoris more than 1 month and had no significant changes in the degree, frequency, nature and inducing factors of angina pectoris
* The severity of angina pectoris of the Canadian Cardiovascular Society (CCS) was classified as Grade I to Grade III, and angina pectoris occurred more than twice a week
* The syndrome differentiation of TCM is Qi stagnation and blood stasis syndrome
* Age ranges from 30 to 79 years old
* Sign the informed consent

Exclusion Criteria:

* Severe cardiopulmonary insufficiency (grade III, IV, severe abnormal pulmonary function);
* Poor control of hypertension (systolic blood pressure (> 160 mmHg) or diastolic blood pressure (> 100 mmHg) after treatment;
* Complicated with liver and kidney function damage, ALT, AST (> 1.5 times of the upper limit of normal value), or Cr (> the upper limit of normal value), combined with hematopoietic system and other serious primary diseases;
* Acute myocardial infarction within 3 months after interventional therapy;
* Cardiac pacemaker;
* Pregnancy, lactation or pregnancy planners;
* Anaphylactic constitution or allergic to known ingredients of research drugs;
* Chest pain caused by other causes (moderate anemia, hyperthyroidism, etc.)
* Those who participated in other clinical drug trials within one month;
* According to the judgement of the researchers, it is not advisable to participate in clinical researchers.
* Other factors affecting ST-T changes in ECG, such as myocardial hypertrophy, left bundle branch block, etc.

Ages: 30 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2018-05-15 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
the changes of curative effect of angina pectoris symptoms | Visit1:introduction period,-14±2days; Visit2:treatment period,-4~0day; Visit3:treatment period,4weeks±4days; Visit4:treatment period,8weeks±4days; Visit5:treatment period, 12weeks±4days
  The number of angina attacks, duration, degree of pain, and the dosage of nitroglycerin are used as indicators for scoring. Score ranges 0-15, the higher the score, the more severe the angina.

SECONDARY OUTCOMES:
Therapeutic effect of TCM syndromes | Visit1:introduction period,-14±2days; Visit2:treatment period,-4~0day; Visit3:treatment period,4weeks±4days; Visit4:treatment period,8weeks±4days; Visit5:treatment period, 12weeks±4days
  The main symptoms of Qi stagnation and blood stasis syndrome are chest pain, chest tightness, secondary symptoms such as palpitation, shortness of breath, chest swelling, fatigue, dark lips, dizziness, veins at the base of tongue, irritability, etc. The severity and presence of these symptoms are used as criteria for scoring. Score ranges 0-28.The higher the score, the more serious it is.
Grading changes of severity of angina pectoris | Visit1:introduction period,-14±2days; Visit2:treatment period,-4~0day; Visit3:treatment period,4weeks±4days; Visit4:treatment period,8weeks±4days; Visit5:treatment period, 12weeks±4days
  Reference to Canadian Cardiovascular Society (CCS) Angina Severity Classification Standard。Ⅰ：General physical activity does not cause angina pectoris, such as walking and going upstairs, but tension, rapid or sustained exertion can cause the onset of angina pectoris.Ⅱ：Daily physical activity is slightly restricted. Walking fast or upstairs, climbing high, walking after meals or upstairs, walking in cold or wind, and emotional excitement can cause angina or only occur within a few hours after waking up. It is limited to walk more than 200 meters or climb stairs above one floor at normal speed.Ⅲ：Daily physical activity is obviously limited, and angina pectoris can occur when walking 100-200 m at normal speed or climbing a staircase.Ⅳ：Angina symptoms can occur when you are slightly active or at rest.
Changes in the number of angina attacks per week | through study completion, an average of 14 weeks
  Frequency of angina pectoris episodes per week
Nitroglycerin dosage | through study completion, an average of 14 weeks
  basic treatment
Seattle Angina Questionnaire,SAQ | Visit1:introduction period,-14±2days; Visit2:treatment period,-4~0day; Visit3:treatment period,4weeks±4days; Visit4:treatment period,8weeks±4days; Visit5:treatment period, 12weeks±4days
  The Seattle Angina Questionnaire (SAQ) measured a total of L9 problems,including physical activity limitation, stable state of angina, frequency of angina attack, satisfaction with treatment, and knowledge of disease. A kind of Assessment of Seattle Scale: The Seattle Angina Scale was divided into 5 items and 19 items: Physical Activity Restriction (PL, Question 1), Angina Stable State (AS, Question 2), Angina Attack (AF, Question 3-4), Treatment Satisfaction (TS, Question 5-8), Disease Cognition (DS, Question 9-11), 19 items of 5 items and the total score of SAQ. The formula is transformed into standard integral, standard integral = (actual score - the lowest score in this respect) / (the highest score in this respect - the lowest score in this respect) * 100, the higher the score, the better the quality of life and the state of body function of patients.
Blood homocysteine | visti1:treatment period,-4~0day; Visit2:treatment period,12weeks±4days
  The changes of blood HCY before and after treatment are compared between the two groups.
Incidence of cardiovascular events | Visit1:treatment period,-4~0day; Visit2:treatment period,4weeks±4days; Visit3:treatment period,8weeks±4days; Visit4:treatment period, 12weeks±4days
  Sudden cardiac death, acute myocardial infarction, heart failure, percutaneous transluminal coronary angioplasty, coronary artery bypass grafting, malignant arrhythmia, cardiogenic cerebrovascular accident, angina pectoris requiring hospitalization, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Fengqin Xu, Doctor, Principal Investigator — Xiyuan Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Xiyuan Hospital, Chinese Academy of Traditional Chinese Medicine, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zhao JN, Zhang Y, Lan X, Chen Y, Li J, Zhang P, Wu LQ, Jia ST, Liu Y, Xu FQ. Efficacy and safety of Xinnaoning capsule in treating chronic stable angina (qi stagnation and blood stasis syndrome): Study protocol for a multicenter, randomized, double-blind, placebo-controlled trial. Medicine (Baltimore). 2019 Aug;98(31):e16539. doi: 10.1097/MD.0000000000016539. PMID 31374015

DOCUMENTS (2):
  • Study Protocol (2018-01-26): https://cdn.clinicaltrials.gov/large-docs/31/NCT03914131/Prot_000.pdf
  • Informed Consent Form (2018-01-26): https://cdn.clinicaltrials.gov/large-docs/31/NCT03914131/ICF_001.pdf